CLINICAL TRIAL: NCT01504633
Title: Can NUtrigenomics / Nutrigenetics Help Explain the Mixed Results on Effect of LCPUFA (DHA) and Iron on Child COgnition?
Brief Title: Nutrigenomics, PUFA, Iron and Cognition Amongst Under-two-year-old Indonesian Children
Acronym: NUPICO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Collaborators: Wageningen University (Other)
Responsible Party: Principal Investigator, Umi Fahmida, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Quadruple
Other Study IDs: NUPICO-Indonesia
Record Dates: First submitted 2011-12-31; First posted 2012-01-05 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Cognitive Ability, General
Keywords: cognitive function; omega-3 PUFA (DHA); iron; nutrigenomics; under-two year old children; Indonesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- DHA+EPA Group (Experimental): DHA/EPA capsule (100mg DHA + 20mg) and placebo syrup per day
  Interventions: Dietary Supplement: DHA/EPA and iron supplementation
- Fe Group (Experimental): Placebo capsule and Fe syrup (16mg elemental iron) per day
  Interventions: Dietary Supplement: DHA/EPA and iron supplementation
- DHA/EPA+Fe Group (Experimental): DHA/EPA capsule (100mg DHA + 20mg) and Fe syrup (16mg elemental iron) per day
  Interventions: Dietary Supplement: DHA/EPA and iron supplementation
- Placebo Group (Experimental): Placebo capsule and placebo syrup
  Interventions: Dietary Supplement: DHA/EPA and iron supplementation

INTERVENTIONS:
Dietary Supplement: DHA/EPA and iron supplementation — 24-week supplementation consisting of daily dosage of DHA/EPA or placebo capsule and iron/placebo syrup Capsule: DHA/EPA (100mg DHA + 20mg per day) or placebo Syrup: Fe syrup (16mg elemental iron per day) or placebo

SUMMARY:
Rationale: Review on the positive effect of long chain polyunsaturated fatty acids (LCPUFA), especially docosahexanoic acid (DHA), supplementation on cognitive function in human using randomized controlled trials (RCTs) showed that results in RCTs were mixed and inconsistent. It has been suggested that the effect may be subtle, which is currently difficult to detect, but could be significant, or there may be individual variation which mediate the effect.

Objectives: This study aims to assess gene-nutrient inter-relation in explaining the effect of LCPUFAs i.e. DHA and/or iron on cognitive functioning of children <24mo in Indonesia. Specifically the study's objectives are: (1) to assess effect of LCPUFA (as DHA oil) and iron (as iron supplement) in altering gene expressions, and (2) to assess the mediating effect of genes involved in fatty acid and iron metabolism in improving serum LCPUFA, alpha-linolenic acids (ALA), DHA and cognitive function.

Study design and study population: The study is a double-blind randomized controlled trial with children aged less than 24 months (window of opportunity). The study area is in East Lombok district, in West Nusa Tenggara province, Indonesia where nutrient intake including iron and presumably LCPUFA, is not optimal.

Intervention: The study is an intervention study, consisting of four groups: DHA, iron, DHA+iron, and placebo (60 subjects/group = 240 subjects in total). Capsule containing 100mg/d DHA or its placebo and syrup containing 16mg/d iron will be given daily for 24 weeks. Before and after the intervention child cognition (as Bayley Mental Developmental Index or MDI score), serum PUFA level, iron status (haemoglobin, transferrin receptor, ferritin), inflammation status (CRP, AGP), gene expression profiles, and potential confounders of child cognition such as lengt-for-age, weight-for-length, and weight-for-age Z-scores, stimulation/home environment, maternal characteristics will be collected.

Study outcome: The primary study outcomes will be cognitive score (as Bayley Mental Developmental Index or MDI score) and gene expression profiles. Secondary study outcomes will be serum PUFA level, iron status (haemoglobin, TfR, ferritin).

Nature and extent of the burden and risks benefit and group relatedness:

Subjects, who will be included into the study will invest 14 hours. The consumption of iron is not associated with any increased risk of iron overload both for infectious (including malaria) and chronic diseases nor consumption of n-3 fatty acids EPA and DHA exceed the US Food and Drug Administrator (FDA) Generally Recognized as Save (GRAS) limit. Venous blood of 5 mL will be drawn at baseline and endline. During screening, children with severe anaemia (Hb<70g/L) will be excluded from the study and referred to the local public health center for further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 12 to 17months old
* Both father and mother of Sasak ethnicity
* Currently breastfed

Exclusion Criteria:

* Birth weight <2500 grams (LBW)
* Congenital malformation and/or disorder that interfered with adequate functioning in daily life
* Hemoglobin value below 70 g/L
* Malaria
* Maternal depression

Ages: 12 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
change in cognitive function (MDI score) | within 24 weeks after start of intervention
  Mental Developmental Index (MDI) score of Bayley Scale of Infant Development (BSID)

CONTACTS AND LOCATIONS:
Overall Officials: Umi Fahmida, PhD, Principal Investigator — SEAMEO Regional Center for Food and Nutrition (RECFON) University of Indonesia
Locations (1):
- SEAMEO Regional Center for Food and Nutrition (RECFON) University of Indonesia, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Arterburn LM, Hall EB, Oken H. Distribution, interconversion, and dose response of n-3 fatty acids in humans. Am J Clin Nutr. 2006 Jun;83(6 Suppl):1467S-1476S. doi: 10.1093/ajcn/83.6.1467S. PMID 16841856
- [Background] Bouwens M, van de Rest O, Dellschaft N, Bromhaar MG, de Groot LC, Geleijnse JM, Muller M, Afman LA. Fish-oil supplementation induces antiinflammatory gene expression profiles in human blood mononuclear cells. Am J Clin Nutr. 2009 Aug;90(2):415-24. doi: 10.3945/ajcn.2009.27680. Epub 2009 Jun 10. PMID 19515734
- [Background] Bouwens M, Grootte Bromhaar M, Jansen J, Muller M, Afman LA. Postprandial dietary lipid-specific effects on human peripheral blood mononuclear cell gene expression profiles. Am J Clin Nutr. 2010 Jan;91(1):208-17. doi: 10.3945/ajcn.2009.28586. Epub 2009 Nov 18. PMID 19923369
- [Background] Cunnane SC, McAdoo KR. Iron intake influences essential fatty acid and lipid composition of rat plasma and erythrocytes. J Nutr. 1987 Sep;117(9):1514-9. doi: 10.1093/jn/117.9.1514. PMID 3116180
- [Background] El-khayat H, Shaaban S, Emam EK, Elwakkad A. Cognitive functions in protein-energy malnutrition: in relation to long chain-polyunsaturated fatty acids. Pak J Biol Sci. 2007 Jun 1;10(11):1773-81. doi: 10.3923/pjbs.2007.1773.1781. PMID 19086537
- [Background] Idjradinata P, Pollitt E. Reversal of developmental delays in iron-deficient anaemic infants treated with iron. Lancet. 1993 Jan 2;341(8836):1-4. doi: 10.1016/0140-6736(93)92477-b. PMID 7678046
- [Background] Koletzko B, Demmelmair H, Schaeffer L, Illig T, Heinrich J. Genetically determined variation in polyunsaturated fatty acid metabolism may result in different dietary requirements. Nestle Nutr Workshop Ser Pediatr Program. 2008;62:35-44; discussion 44-9. doi: 10.1159/000146246. PMID 18626191
- [Background] Kwik-Uribe CL, Gietzen D, German JB, Golub MS, Keen CL. Chronic marginal iron intakes during early development in mice result in persistent changes in dopamine metabolism and myelin composition. J Nutr. 2000 Nov;130(11):2821-30. doi: 10.1093/jn/130.11.2821. PMID 11053527
- [Background] McCann JC, Ames BN. Is docosahexaenoic acid, an n-3 long-chain polyunsaturated fatty acid, required for development of normal brain function? An overview of evidence from cognitive and behavioral tests in humans and animals. Am J Clin Nutr. 2005 Aug;82(2):281-95. doi: 10.1093/ajcn.82.2.281. PMID 16087970
- [Background] McCann JC, Ames BN. An overview of evidence for a causal relation between iron deficiency during development and deficits in cognitive or behavioral function. Am J Clin Nutr. 2007 Apr;85(4):931-45. doi: 10.1093/ajcn/85.4.931. PMID 17413089
- [Background] Murray-Kolb LE, Beard JL. Iron deficiency and child and maternal health. Am J Clin Nutr. 2009 Mar;89(3):946S-950S. doi: 10.3945/ajcn.2008.26692D. Epub 2009 Jan 21. PMID 19158210
- [Background] Oloyede OB, Folayan AT, Odutuga AA. Effects of low-iron status and deficiency of essential fatty acids on some biochemical constituents of rat brain. Biochem Int. 1992 Aug;27(5):913-22. PMID 1417923
- [Background] Smuts CM, Tichelaar HY, van Jaarsveld PJ, Badenhorst CJ, Kruger M, Laubscher R, Mansvelt EP, Benade AJ. The effect of iron fortification on the fatty acid composition of plasma and erythrocyte membranes in primary school children with and without iron deficiency. Prostaglandins Leukot Essent Fatty Acids. 1995 Jan;52(1):59-67. doi: 10.1016/0952-3278(95)90098-5. PMID 7708822
- [Background] Stangl GI, Kirchgessner M. Different degrees of moderate iron deficiency modulate lipid metabolism of rats. Lipids. 1998 Sep;33(9):889-95. doi: 10.1007/s11745-998-0285-8. PMID 9778136
- [Background] Rajilic-Stojanovic M, Heilig HG, Molenaar D, Kajander K, Surakka A, Smidt H, de Vos WM. Development and application of the human intestinal tract chip, a phylogenetic microarray: analysis of universally conserved phylotypes in the abundant microbiota of young and elderly adults. Environ Microbiol. 2009 Jul;11(7):1736-51. doi: 10.1111/j.1462-2920.2009.01900.x. Epub 2009 Mar 11. PMID 19508560
- [Derived] Shinta D; Asmarinah; Adhiyanto C, Htet MK, Fahmida U. The Association of TMPRSS6 Gene Polymorphism and Iron Intake with Iron Status among Under-Two-Year-Old Children in Lombok, Indonesia. Nutrients. 2019 Apr 19;11(4):878. doi: 10.3390/nu11040878. PMID 31010126
- [Derived] Fahmida U, Htet MK, Adhiyanto C, Kolopaking R, Yudisti MA, Maududi A, Suryandari DA, Dillon D, Afman L, Muller M. Genetic variants of FADS gene cluster, plasma LC-PUFA levels and the association with cognitive function of under-two-year-old Sasaknese Indonesian children. Asia Pac J Clin Nutr. 2015;24(2):323-8. doi: 10.6133/apjcn.2015.24.2.17. PMID 26078250
- See also: South East Asia Ministers of Education Organization, Regional Center for Food and Nutrition, University of Indonesia — http://seameo-recfon.org/